CLINICAL TRIAL: NCT06730854
Title: Association Between Elevated Liver Functions Tests Following Cardiac Surgery and Acute Kidney Injury - a Restrospectiv Single Center Cohort Study
Brief Title: Association Between Liver Function Tests and Acute Kidney Injury in Cardiac Surgery Patients
Acronym: TransAKI
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2024-0453
Record Dates: First submitted 2024-11-26; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Cardiac Surgery Associated - Acute Kidney Injury; Acute Kidney Injury
Keywords: liver enzymes; acute kidney injury; cardiac surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Main cohort of patient: In the included patients the occurrence of acute kidney injury (AKI) will be investigated. So patient will be grouped as 'no AKI' and 'AKI' For the subanalysis, patient will be grouped according to their admission central venous pressure.
  There are no interventions.

SUMMARY:
A sudden decline in function of the kidneys is a common problem that can happen after heart surgery. It can have serious effects on a patient's recovery and long-term health, potentially leading to permanent kidney problems or heart-related issues. One of the main reasons kidney problems occurs is due to changes in blood flow caused by the heart not pumping well enough. These changes may harm the kidneys, but other organs as well such as the liver.

This study aims to find out if there is a relationship between elevated levels of liver function blood tests and the decline in kidney function.

DETAILED DESCRIPTION:
In this study data will be retrospectively collected from the intensive care patient management system for patients admitted postoperatively to the cardiac intensive care unit (ICU) following cardiac surgery. The inclusion period spans from 2012 to 2017 (5 years) and includes about 3,500 patients.

For all included patients, retrospective data collection will include variables related to renal function, fluid balance, hemodynamics, and transaminase levels. Additionally, demographic information, surgical procedure details, comorbidities, and laboratory values will be gathered.

Cardiac surgery-associated acute kidney injury (CSA-AKI) has a multifactorial etiology influenced by non-modifiable factors such as age, comorbidities (e.g., heart failure/ejection fraction, chronic kidney disease, hypertension, diabetes), medication use (NSAIDs, ACE inhibitors/ARBs), type of surgery, duration of surgery/cardiopulmonary bypass time. Central venous pressure (CVP) can serve as a marker of venous congestion, which may contribute to the development of AKI. Venous congestion may also result in elevated transaminase levels.

The primary aim of this study is to investigate the association between postoperative transaminase elevation in the ICU and the development of AKI during the intensive care stay. Data about transaminases will be collected in the first 24 hours after ICU admission. The occurrence of AKI and its severity will be investigated within 72 hours after cardiac surgery. Furthermore, the relationship between the transaminase elevation and the severity of acute kidney injury will be examined, as well as the association between central venous presure (CVP) and transaminase levels postoperatively in the ICU.

Acute kidney injury will be defined according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria, with severity classified based on the KDIGO staging system.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* admission on intensive care after cardiac surgery
* available data about liver enzymes

Exclusion Criteria:

* chronic kidney disease with (estimated) glomerular filtration rate below 30mL/min/1.73 m2 or renal replacement therapy (RRT) dependent
* patient on extracorporal membrane oxygenator (ECMO) before or after cardiac surgery
* patient with or planned surgery for Left ventricular assist device (LVAD)
* inotropics or vasopressore before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cardiac surgery patients screened for eligibility were admitted on the cardiac surgery intensive care unit of Ghent University hospital between 1 Januari 2012 until 31 december 2017
Sampling Method: Non-Probability Sample
Enrollment: 3415 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Association between liver enzymes and acute kidney injury | Data about liver enzymes will be collected at ICU admission, and 12 hours and 24 hours after ICU admission. The occurrence of acute kidney injury within 72 hours after ICU admission will be investigated
  Investigation of the association between liver enzymes (alanine aminotransferase (AST); aspartate aminotransferase (ALT)) and development of acute kidney injury. Data about liver enzymes will be collected at ICU admission, and 12 hours and 24 hours after ICU admission. AKI is defined by the Kidney Disease Improving global outcome definition by using both the serum creatinine and urine output criteria.

SECONDARY OUTCOMES:
Association between liver enzymes and the severity of acute kidney injury | Data about liver enzymes will be collected at ICU admission, and 12 hours and 24 hours after ICU admission. The occurrence of the different severity stages of acute kidney injury within 72 hours after ICU admission will be investigated
  Investigation of the association between liver enzymes (alanine aminotransferase (AST); aspartate aminotransferase (ALT)) and the sevirity of the developed acute kidney injury. AKI severity is defined by the Kidney Disease Improving global outcome (KDIGO) classification: stage 1, stage 2 and stage 3. Stage 3 is the most severe form of kidney injury, including the use of renal replacement therapy (RRT)
association of central venous pressure with elevated liver enzymes and acute kidney injury | Data about central venous pressure will be collected during the first 24 hours after ICU admission.
  Investigation of the association between elevated central venous pressure and elevation in liver enzymes (alanine aminotransferase (AST); aspartate aminotransferase (ALT)) and the development of acute kidney injury (severity)

CONTACTS AND LOCATIONS:
Overall Officials: Wim Vandenberghe, MD; PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent university hospital, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No
Due to European Data Protection regulation, no individual participant data will be shared, only the analysed data.